CLINICAL TRIAL: NCT05728606
Title: Robot-assisted D2 Distal Gastrectomy Following Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE-03
Record Dates: First submitted 2023-01-20; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted D2 distal gastrectomy (Experimental): Robot-assisted D2 distal gastrectomy after 3-Cycle SOX neoadjuvant chemotherapy
  Interventions: Procedure: Robot-assisted D2 distal gastrectomy

INTERVENTIONS:
Procedure: Robot-assisted D2 distal gastrectomy — Robot-assisted D2 distal gastrectomy after 3-Cycle SOX neoadjuvant chemotherapy

SUMMARY:
To evaluate the safety of robot-assisted radical gastrectomy with D2 lymph node dissection in postoperative complications in patients with neoadjuvant chemotherapy for gastric cancer (cT3-4a, N+, M0).

ELIGIBILITY:
Inclusion Criteria:

Age from over 18 to under 75 years; Primary gastric adenocarcinoma (including pap, tub, muc, sig, and por) confirmed pathologically by endoscopic biopsy; cT3-4a, N-/+, M0 according to the AJCC 8th Cancer Staging Manual; Without peritoneal metastasis (examined by laparoscopic examination); Radical resection (R0) through distal subtotal gastrectomy with D2 lymphadenectomy is anticipated; Performance status 0 or 1 (Eastern Cooperative Oncology Group) ; ASA (American Society of Anesthesiology) score ≤ 3;

Normal hemodynamic indices:

Blood cell count: HB ≥ 90g/L, ANC ≥ 1.5×109/L, PLT ≥ 80×109/L; Liver and renal function: BIL<1.5 times of the upper limit of normal reference values, ALT and AST<2.5 times of the upper limit of normal reference values, and Crea≤1 time of upper limits of normal reference values.

Therapeutic response rating after neoadjuvant chemotherapy is CR, PR, SD, or Therapeutic response rating after neoadjuvant chemotherapy is PD, tumor is expected to have radical resection; Subjects are still willing to continue participating in this clinical trial.

Exclusion Criteria:

History of upper abdominal surgery (include endoscopic mucosal resection or endoscopic submucosal dissection, except for laparoscopic cholecystectomy); History of acute pancreatitis; Enlarged or bulky regional lymph node (diameter>3cm) by imaging exam; Patients have received neoadjuvant therapy prior to screen work; History of other malignant disease within the past five years; History of cerebrovascular accident within the past six months; History of continuous systematic administration of corticosteroids within the past month; Scheduled simultaneous surgery for other disease; Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer; Pyloric obstruction; FEV1<50% of predicted value; Women who are pregnant or lactating at the time of screening; Severe mental disorder; Participating in other clinical studies; Refused to sign the informed consent;

Therapeutic response rating after neoadjuvant chemotherapy is PD, involvement of adjacent structures(T4b), distal metastasis(M1), or enlarged or bulky regional lymph node (diameter>3cm) by preoperative imaging Patients cannot complete 3 cycles of chemotherapy due to intolerance; After 3 cycles of neoadjuvant chemotherapy, patients cannot tolerate surgery due to severe adverse reactions, or ASA score ≥ 4 ; Patients undertake emergency operation due to tumor bleeding, perforation or obstruction during chemotherapy; After signing the informed consent, the patient withdraws from this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Total incidence of postoperative complications | Postoperative 30 days
  Postoperative complications are defined as complications occurring within 30 days after surgery, and will be classified according to the Clavien-Dindo classification system

SECONDARY OUTCOMES:
Hospital mortality | Postoperative 30 days
  Hospital mortality is defined as death occurring within 30 days after initial surgery, regardless of the cause
R0 resection rate | The day of surgery
Robotic surgical completion rate | The day of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei, China